CLINICAL TRIAL: NCT05587153
Title: Comparative Study Between the Perfusion Index and Positional Haemodynamic Changes for Prediction of Hypotension After Spinal Anaesthesia in Caesarean Section
Brief Title: Perfusion Index vs Positional Hemodynamic Changes to Predict Hypotension After Spinal Anaesthesia in Caesarean Section
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Other Study IDs: 9293/2-2-2022
Record Dates: First submitted 2022-03-08; First posted 2022-10-19 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Post Spinal Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational study in parturient who will be recruited for the study: this study will include the eligible parturient who will be assessed by perfusion index and by positional hemodynamic changes.
  Interventions: Other: perfusion index in all parturient recruited for the study

INTERVENTIONS:
Other: perfusion index in all parturient recruited for the study — Using perfusion index and positional hemodynamic changes for the prediction of postspinal hypotension in all parturient recruited for the study
  Other Names: positional haemodynamic changes between supine and right lateral position in parturient .

SUMMARY:
Comparative Study between the Perfusion Index and Positional Haemodynamic Changes for Prediction of Hypotension after Spinal Anaesthesia in Caesarean Section

DETAILED DESCRIPTION:
Hypotension following spinal anaesthesia may cause maternal dizziness, nausea, vomiting and fetal acidosis, administration of prophylactic vasopressor agents in pregnant women may cause undesirable effects on the mother and fetus. Perfusion index is the ratio of a pulsatile to a non-pulsatile fraction of blood volume. The increase of the pulsatile fraction manifested during vasodilatation corresponds to a higher PI. So, the patients with a higher PI have a higher risk for post-spinal hypotension. Elevated sympathetic activity before neuraxial anaesthesia was associated with a higher risk for post-spinal hypotension. The significant variability in haemodynamic after the positional change indicates higher sympathetic activity. The high the rise in autonomic activity, the higher the risk for post-spinal hypotension

AIM OF THE WORK:

Prediction of hypotension after spinal anaesthesia in caesarean section either by perfusion index and positional haemodynamic changes

Grouping:

All the recruited patients will be assessed by perfusion index. and by positional haemodynamic changes

ELIGIBILITY:
Inclusion criteria

* Parturient acceptance.
* American Society of Anesthesiologists (ASA) II
* arturient with be gestational age >36 weeks and <41 weeks.
* Body mass index (BMI) ≤35kg/m2
* elective caesarean section delivery

Exclusion criteria

* preeclampsia
* eclampsia,
* gestational diabetes
* Contraindication to regional anaesthesia as allergy, coagulation abnormalities or infection in site of injection.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant female patients above 18 years who will undergo cesarean section
Study Population: Pregnant women undergoing an elective caesarean section delivery.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Prediction of post-spinal hypotension using PI | 6 months
  To correlate between perfusion index and hypotension after spinal anaesthesia in caesarean section

SECONDARY OUTCOMES:
Prediction of post-spinal hypotension using positional hemodynamic changes | 6 months
  To correlate between positional haemodynamic changes and hypotension after spinal anaesthesia in caesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa Abdelhaleem, MD, Study Director — Faculty of medicine, Zagazig University Hospitals
Locations (2):
- Egypt (2):
  - Faculty of medicine, Zagazig
  - Ramy, Zagazig

IPD SHARING:
Plan to Share IPD: Undecided